CLINICAL TRIAL: NCT03431298
Title: The Benefit of Increasing Physical Activity and Functional Movement Control for Patients With Stage II or III Knee Osteoarthritis
Brief Title: The Benefit of Functional Movement Control for Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-M03-038
Record Dates: First submitted 2018-01-28; First posted 2018-02-13 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Physical activity; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise & movement control (Experimental): The duration of intervention is 8 weeks.
  * Individualized functional movement control training is 60 min/week
  * Aerobic exercise is 60 min/week
  Interventions: Behavioral: Aerobic exercise & movement control
- Aerobic exercise (Active Comparator): The duration of intervention is 8 weeks.
  * Frequency: 2 times/ week
  * Duration: 60min/ time
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise & movement control — The aerobic exercise content is no different between the experimental group and the active comparator group.
  The movement control is individual training which divided into fourths progressing sessions.
  * First, lumbo-pelvic and hip dynamic direction control.
  * Second, trunk muscle groups, hip muscle groups and thigh muscle groups extensibility control.
  * Third, trunk muscle groups and hip muscle groups through range control.
  * Fourth, functional movement control training
  Arms: Aerobic exercise & movement control
Behavioral: Aerobic exercise — The aerobic exercise will organized in groups. Each group has 6-8 persons. The exercise form is fixed at each time.
  The description of exercise form is as below:
  * 10 min Warm up
  * 40 min Aerobic exercise (which focus on lower extremity muscle strengthening and increasing muscle endurance)
  * 10 min Cool down
  Arms: Aerobic exercise

SUMMARY:
The study purpose is to explore the effect of functional movement control for patients who have stage II or III degenerative knee joint disease and also physical inactive. Half of patients will receive aerobic exercise and functional movement control training in combination, while the other will simply receive aerobic exercise.

DETAILED DESCRIPTION:
Physical inactivity, which is a common phenomenon among patients with degenerative knee joint disease has been proved a predictor of increased symptoms and poor general health. However, changing the lifestyle of people with this disease who is physical inactive is still a problem which has not been solved. Knee pain may act as barrier to engage in physical activity and can influence patient's movement performance.

The different effectiveness between the aerobic exercise and functional movement control training.

Aerobic exercise has been proved could improve knee pain for the patients with degenerative knee joint disease.

The functional movement control training could improve knee alignment during walking and other functional activities to increase patient's movement awareness.

ELIGIBILITY:
Inclusion Criteria:

* Participant who was diagnosed has knee osteoarthritis
* Above 40 years old
* Participant who didn't achieve at least 150 min moderate intensity physical activity level per week

Exclusion Criteria:

* Patients with walking disability
* Cannot complete 8 weeks intervention program
* Received arthroscopy or other surgery before 6 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
reaching proportions of the level of health enhancing physical activity | up to 6 months after intervention
  the recommended level of health enhancing physical activity is at least 150 min of moderate intensity physical activity per week

SECONDARY OUTCOMES:
Partial foot pressure as a percentage of body weight | Baseline and up to 1 week after intervention
  The area footprinted during gait was divided into 6 parts according to the average foot areas of subject. Then, the partial foot pressure as a percentage of body weight was calculated as the average value during the stance phase of each step in each part as a percentage of the body weight.
Partial foot area as a percentage of body mass index | Baseline and up to 1 week after intervention
  The area footprinted during gait was divided into 6 parts. The partial foot area as a percentage of body mass index was calculated as the average value during the stance phase of each step in each part as a percentage of the body mass index.
Gait Cadence | Baseline and up to 1 week after intervention
  the number of steps per minute
Walking speed | Baseline and up to 1 week after intervention
  the velocity of single step
Single leg stance time | Baseline and up to 1 week after intervention
  the time of the stance phase of each foot
Step length | Baseline and up to 1 week after intervention
  the distance between the first point of contact of a limb with the ground and the first point of contact of the limb on the opposite side
Step width | Baseline and up to 1 week after intervention
  the distance between the centre of the first heel contact and the following one calculated perpendicularly to the direction of the horizontal axis drawn between the feet
Axis angle | Baseline and up to 1 week after intervention
  the angle formed by the medial tangent of the foot and the line from the second/third toe to the center of the heel
The Knee injury and Osteoarthritis Outcome Score | Baseline and up to 1 week after intervention
  A questionnaire to assess the patient's opinion about their knee and associated problems.
Sort Form-12v2 Healthy Survey | Baseline and 1, 3, 6 month after intervention
  12 question to measure functional health and well-being from the patient's point of view

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yin Chen, PhD, Principal Investigator — National Yang-Ming University The Department of Physical Therapy and Assistive Technology
Locations (1):
- Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No